CLINICAL TRIAL: NCT06504277
Title: A Randomized Controlled Trial (RCT) Comparing the Effect of Low Versus Standard Pressure Pneumoperitoneum on Post-operative Shoulder Tip Pain in Patients Undergoing Laparoscopic Gynecologic Surgery for Benign Indications
Brief Title: Low Versus Standard Pressure Pneumoperitoneum on Shoulder Tip Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Women's College Hospital (Other)
Responsible Party: Principal Investigator, Mara Sobel, Associate Professor, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-0008-E
Record Dates: First submitted 2024-07-04; First posted 2024-07-16 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Surgery; Laparoscopic; Laparoscopy; Penumoperitoneum; Post-operative Pain; Post-operative Recovery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This proposed study is a single-center parallel group RCT comparing the use of low (10 mm Hg) versus standard pressure (15 mm Hg) pneumoperitoneum at the time of benign gynecologic laparoscopic surgery. Participants will be selected using a convenience sample from Women's College Hospital operating room list. All potentially eligible patients will be invited to participate in this study by the MIS fellow on the day of surgery up to 2 hours before the scheduled surgery.
  We will create a randomization list in equal ratio with study numbers 1 to 82. A member of the research team who will have no interaction with patients in this study will prepare the low and standard pressure envelopes and label them according to the randomization list.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study participants will be randomized on the day of surgery, and the research nurse will set the insufflation pressure to the pre-randomized pressure identified in the envelope. The surgeon, research team, participants and data analysts will be blinded to treatment group.
  Study participants will be randomized on the day of surgery. After Veress-needle insufflation and laparoscopic port insertion at a pneumoperitoneum of 20mmHg (standard entry pressure), the patient will be placed in Trendelenberg position. At this time, the research nurse will set the insufflation pressure to the pre-set randomized number. This insufflation pressure will be blinded on the machine from the surgeon. If the surgeon is not satisfied with the visibility, they may ask to set the pressure to 15mmHg, however, they will remain blinded. The surgeon, research team, participants and data analysts will be blinded to treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Pressure (Active Comparator): Patients undergoing laparosocpy at standard pressure (15 mm Hg)
  Interventions: Other: Standard Pressure Group (No intervention- active comparator)
- Low Pressure (Experimental): Patients undergoing experimental intervention of low pressure pneumoperitoneum (10 mm Hg)
  Interventions: Procedure: Low Pressure Penumoperitoneum

INTERVENTIONS:
Procedure: Low Pressure Penumoperitoneum — Maintained Pneumoperitoneum with low pressure of 10 mm Hg
  Arms: Low Pressure
Other: Standard Pressure Group (No intervention- active comparator) — Maintained Pneumoperitoneum at standard pressure of 15 mm Hg
  Arms: Standard Pressure

SUMMARY:
This proposed study is a single-center, double blind, parallel group RCT comparing the use of low (10 mm Hg) versus standard pressure (15 mm Hg) pneumoperitoneum at the time of benign gynecologic laparoscopic surgery. Patients will be randomized to the control group (standard pressure) or the intervention group (low pressure) and surgeons will be blinded to the study pressure. Data on post-operative recovery and pain scores will be recorded for each patient.

DETAILED DESCRIPTION:
Primary Objective: The primary objective of this study is to determine the effect of low (10 mm Hg) versus standard pressure (15 mm Hg) pneumoperitoneum on post-operative shoulder pain on post operative day one following laparoscopic gynecologic surgery for benign indication.

Secondary Objective: Secondary outcomes measured will include post-operative shoulder tip pain at 1 and 2 hours, QoR score (Appendix A) on POD 1, incidence of post-operative shoulder tip pain (defined as pain rating above zero) at 1, 2, and POD 1, generalized pain, nausea and bloating at 1 and 2 hours and POD 1, as well as rescue analgesia consumption before discharge and use up to POD1. The investigators will also measure intraoperative time, complication rates, estimated blood loss, surgeon visibility rating and anesthetist satisfaction rating, and time to patient discharge. Additionally, investigators will assess rate of failure to complete the surgery at designated pressure (i.e. request to increase pressure).

This proposed study is a single-center parallel group RCT comparing the use of low (10 mm Hg) versus standard pressure (15 mm Hg) pneumoperitoneum at the time of benign gynecologic laparoscopic surgery. Participants will be selected using a convenience sample from Women's College Hospital operating room list. All potentially eligible patients will be invited to participate in this study by the MIS fellow on the day of surgery up to 2 hours before the scheduled surgery. Study consent will be obtained by the MIS fellow or research assistant after the patient has had sufficient time to consider participation in the study.

The investigators will create a randomization list using a computer-generated allocation sequence in equal ratio with study numbers 1 to 82. A member of the research team who will have no interaction with patients in this study will prepare the low and standard pressure envelopes and label them according to the randomization list. Study participants will be randomized on the day of surgery, and the research nurse will set the insufflation pressure to the pre-randomized pressure identified in the envelope. The surgeon, research team, participants and data analysts will be blinded to treatment group. Patients will receive standardized peri-operative care during their operation.

Post-operative pain, nausea, and medication use will be assessed in the PACU. Patients will also be contacted on POD1 to assess post-operative pain scores, calculate total narcotic consumption and elicit any adverse events.

Primary Endpoints: The primary endpoint is post-operative shoulder tip pain measured on POD 1 following surgery by a self-administered NRS for pain. A NRS is a line measuring from 0-10 that rates pain from none (0) to the worst pain imaginable (10). A NRS for subjective pain assessment is a well-established validated measurement tool that has been shown in numerous studies to provide a clinically useful distribution of responses and a detectable treatment effect [Clivatti et al, 2009].

Secondary Endpoints: Secondary outcome measures will include: (a) NRS scores for shoulder-tip pain at 1 and 2 hours (b) QoR score on POD1, (c) NRS scores for generalized pain at 1 and 2 hours and on POD1 (d) post operative nausea, vomiting, and bloating at 1 and 2 hours and on POD1 (e) narcotic consumption measured as total dose of narcotics in PACU and between discharge and the POD1 phone call (f) surgical time (g) estimated blood loss (h) adverse effects/complication rates in hospital and reported by the POD1 phone call (i) surgeon visibility rating and (j) anesthetist satisfaction rating.

ELIGIBILITY:
Inclusion Criteria: The participant must meet all of the inclusion criteria to eligible for this clinical trial:

1. All ages > or = to 18 years old;
2. Must be deemed to have capacity to provide informed consent;
3. Must sign and date the informed consent form;
4. Stated willingness to comply with all study procedures;
5. Must be undergoing unilateral or bilateral salpingo-oopherectomy or salpingectomy or ovarian cystectomy;

Exclusion Criteria: An individual who meets any of the following criteria will be excluded from participation in this clinical trial:

1. Previous midline laparotomy;
2. Gynecological cancer beyond stage 1 disease;
3. Chronic pain;
4. Known diagnosis of endometriosis or evidence of endometriosis intra-operatively;
5. Fibromyalgia;
6. BMI >50;
7. Language barrier;
8. Inability to communicate or provide informed consent;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-07-10 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Shoulder Tip Pain | Post-op day 1
  The primary endpoint is post-operative shoulder tip pain measured on post-op day 1 following surgery by a self-administered NRS (numeric rating score) for pain, on a scale from 0 (no pain) to 10 (worst pain imaginable).

SECONDARY OUTCOMES:
Shoulder Tip Pain (Short-term) | 1 and 2 hours after surgery
  NRS (numeric rating score) scores for shoulder-tip pain at 1 and 2 hours on a scale from 0 (no pain) to 10 (worst pain imaginable)
Quality of Recovery (QoR) score | Post-op day 1
  QoR (Quality of Recovery) score on post-op day 1: a pre-validated score out of 150 (higher score corresponds to better recovery)
Generalized Pain Score | 1, 2 hours post-op and post-op day 1
  Generalized pain at 1 and 2 hours and on post-op day 1. Self-reported NRS pain score on a scale 0-10.
Incidence of Nausea and Vomitting | 1, 2 hours post-op and post-op day 1
  Documented incidence (yes or no) of nausea, vomiting, and bloating at 1 and 2 hours and on post-op day 1. Incidence/presence of nausea and vomiting is worse.
Narcotic use | Post-op day 1
  Narcotic consumption measured as total dose of narcotics in PACU and between discharge and the post-op day1 phone call
Surgical time | Duration of surgery (day surgery)
  Duration of surgery
Estimated blood loss | Duration of surgery (day surgery)
  Estimated blood loss
Adverse Effect/Complications | Post-op day 1
  Adverse effects/complication rates in hospital and reported by post-op day 1 phone call
Surgeon visibility | Duration of surgery
  Surgeon visibility rating: visibility during surgery assessed by surgeon rating on a 5-point Likert scale. Greater score indicates better visibility.
Anesthetist satisfaction | Duration of surgery
  Anesthetist satisfaction rating measured as anesthetist satisfaction with ventilation during surgery. Assessed by anesthetist rating on a 5-point Likert scale (higher score is better).

CONTACTS AND LOCATIONS:
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Undecided